CLINICAL TRIAL: NCT06036420
Title: Flashed Light Therapy for Adolescents With ADHD and Delayed Sleep Timing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Emily J. Ricketts, PhD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-000489
Record Dates: First submitted 2023-05-17; First posted 2023-09-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: ADHD
Keywords: ADHD; light flashes; CBT; sleep
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; photopsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- 1) Flashed Light Therapy, 2) Flashed Light Therapy with Cognitive Behavioral Therapy (Experimental): Treatment Phase 1 (2 weeks duration): light flashes administered for 60 minutes daily beginning 75 minutes prior to the participant's average morning wake time and ending 15 minutes before average morning wake time.
  Treatment Phase 2 (4 weeks duration): will begin immediately following phase 1 and involve daily light flashes (as described above) combined with weekly 50-minute videoconference-delivered cognitive-behavioral therapy.
  Interventions: Device: Flashed Light Therapy; Behavioral: Videoconference-delivered Cognitive Behavioral Therapy

INTERVENTIONS:
Device: Flashed Light Therapy — Light flashes will be presented over 60 minutes as 3-millilisecond flashes of white light at 4,000 lux every 20 seconds
  Other Names: Light flashes
Behavioral: Videoconference-delivered Cognitive Behavioral Therapy — Treatment will involve psychoeducation on sleep, circadian rhythms and light exposure, motivational interviewing, advancing of bedtime schedule, time management and coping with poor sleep, sleep hygiene, stimulus control, sleep restriction, and cognitive restructuring for worry.

SUMMARY:
The primary aim of the present research project is to examine the feasibility, as measured by treatment perceptions, and tolerability, as measured by adherence and attrition, of two weeks of flashed light therapy alone followed by four weeks of daily flashed light therapy combined with four weekly videoconference-delivered cognitive behavioral therapy sessions targeting circadian rhythms and sleep in four adolescents aged 14 to 17 years with attention-deficit/hyperactivity disorder and delayed sleep-wake schedules.

DETAILED DESCRIPTION:
Participation in this research will last about 7 weeks. Participation will involve an initial screening visit lasting 3 hours to assess eligibility. This visit will involve interviews and tasks to assess for psychiatric diagnosis, sleep history, ADHD severity, and thought patterns. Participants and parents will also complete questionnaires assessing parent-reported and self-reported ADHD severity, personal and family demographics, and medical and psychiatric history. Following this visit, participants will be asked to monitor their sleep for 7 nights using a sleep watch and sleep diary, and provide daily report of bedtimes and risetimes via text message.

After sleep monitoring, an 8-hour baseline assessment visit involving interviews, questionnaires, and saliva sampling will be scheduled from 7 hours before average habitual bedtime up until average bedtime to assess the internal body clock. The morning following the baseline assessment, light therapy will begin and continue daily for two weeks. During the two-week period, participants will monitor sleep nightly using a sleep watch and sleep diary.

Following termination of the two-week course of flashed light therapy, participants will complete an 8-hour mid-treatment assessment involving interviews, questionnaires, and saliva sampling, as described above. Following this assessment, participants will begin weekly 50-minute individual videoconference-delivered cognitive behavioral therapy while continuing to use the flashed light therapy device and monitor sleep (via sleep diary, watch, and sleep location verification) for a duration of four weeks. Following treatment, participants will have a post-treatment 8-hour assessment, again involving interviews, questionnaires, and a salivary assessment of the internal body clock, as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 14 to 17 years
2. Current DSM-5 diagnosis of attention-deficit/hyperactivity disorder (any type)
3. Self-reported average bedtime of 11:00 pm or later, with difficulty shifting bedtime earlier and difficulty waking up early enough in the morning
4. Evening chronotype (i.e., score ≤ 27 on the Morningness-Eveningness scale for Children)
5. Clinically significant ADHD severity (ADHD-Rating Scale-5 score ≥ 24)
6. Moderate global functioning impairment or worse (Clinical Global Impression-Severity scale score ≥ 4)
7. Attending school (i.e., standard school year or summer school) during study enrollment
8. Fluency in English

Exclusion Criteria:

1. Current or lifetime diagnosis of bipolar Disorder, psychosis, autism spectrum disorder, or pervasive developmental disorder
2. Alcohol or substance dependence or suicidality within the past 6 months
3. Current depression or anxiety in the severe range or higher
4. Sleep disorder present besides delayed sleep-wake phase disorder (Clinical Sleep History Interview)
5. Sleep solely in the prone position (i.e., on stomach)
6. Full scale IQ ≤ 80 (Wechsler Abbreviated Scale for Intelligence-II)
7. Use of any over-the-counter (e.g., melatonin, Benadryl) or prescribed sleep medication in the past month or planned use during the study
8. Changes to any psychiatric medication within one month of study enrollment or planned changes during the study
9. Use of photosensitizing medication within one month of study enrollment or planned during the study
10. Participation in behavior therapy for sleep and/or ADHD within 3 months of study enrollment or planned participation during the course of the study
11. Use of light therapy within 6 months of study enrollment or planned use during the study
12. Travel across > 2 time zones within one month of study enrollment or planned travel outside of the time zone of participation during the study
13. Structural barriers to sleep (e.g., night shift work, extracurriculars scheduled until late in the evening, early rising for sports practice)
14. Medical or neurological condition (e.g., seizure disorder, chronic migraines) that would interfere in the individual's ability to participate

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Treatment Feasibility: Child-reported | 7 weeks
  Child rating of how acceptable they find the treatment to be on a scale from 1 (very unacceptable) to 7 (very acceptable).
Treatment Feasibility: Parent-reported | 7 weeks
  Parent rating of how acceptable they find the treatment to be on a scale from 1 (very unacceptable) to 7 (very acceptable).
Treatment Tolerability: Treatment Adherence | 7 weeks
  The number of days the participant was exposed to morning light therapy per self-report tracker.
Treatment Tolerability: Attrition | 7 weeks
  The number of participants who withdrew from the study out of the total cases enrolled.

SECONDARY OUTCOMES:
Assessment Tolerability: Child-reported | 7 weeks
  Child rating of how tolerable they find the study assessments to be on a scale from 1 (very intolerable) to 7 (very tolerable).
Assessment Tolerability: Parent-reported | 7 weeks
  Parent rating of how tolerable they find the study assessments to be on a scale from 1 (very intolerable) to 7 (very tolerable).
Treatment Sensitivity of Circadian Phase | 7 weeks
  Change in clock time of dim-light melatonin onset across baseline, mid-treatment, and post-treatment assessment timepoints.
Treatment Sensitivity of Sleep Onset Time | 7 weeks
  Change in clock time of sleep onset across baseline, mid-treatment, and post-treatment assessment timepoints, as measured by actigraphy.
Treatment Sensitivity of Sleep Duration | 7 weeks
  Change in total sleep time (total number of minutes spent asleep during the sleep episode) across baseline, mid-treatment, and post-treatment, as measured by actigraphy.
Treatment Sensitivity of Clinician-rated ADHD Severity (ADHD-RS-5) | 7 weeks
  Change in clinician rated ADHD Rating Scale-5 (ADHD-RS-5) total score across baseline, mid-treatment, and post-treatment assessment timepoints. The ADHD-RS-5 is an 18-item clinical rated scale assessing ADHD symptoms and the extent to which these symptoms exact impairment (DuPaul et al., 2016). Clinicans rate symptom severity and impairment on a scale ranging from 0 (none) to 3 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Ricketts, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Semel Institute for Neuroscience and Human Behavior, University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DuPaul, G. J., Power, T. J., Anastopoulos, A. D., & Reid, R. (2016). ADHD Rating Scale-5 for children and adolescents: Checklists, norms, and clinical interpretation. The Guilford Press.
- [Background] Kaplan KA, Mashash M, Williams R, Batchelder H, Starr-Glass L, Zeitzer JM. Effect of Light Flashes vs Sham Therapy During Sleep With Adjunct Cognitive Behavioral Therapy on Sleep Quality Among Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2019 Sep 4;2(9):e1911944. doi: 10.1001/jamanetworkopen.2019.11944. PMID 31553469